CLINICAL TRIAL: NCT03734978
Title: Division of Neonatology, Zekai Tahir Burak Maternity Teaching Hospital, Clinical Professor
Brief Title: Association Between Different Blood Groups and Sepsis in Preterm Infants
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ufuk Cakir (Other)
Collaborators: Zekai Tahir Burak Women's Health Research and Education Hospital (Other)
Responsible Party: Sponsor-Investigator, Ufuk Cakir, Principal Investigator, Ankara University
Organization: Ankara University (Other)
Other Study IDs: BGaPS
Record Dates: First submitted 2018-11-02; First posted 2018-11-08 (Actual); Last update posted 2018-11-08 (Actual); Status verified 2018-11

CONDITIONS: Blood Group Antigen Abnormality; Prematurity; Sepsis
Keywords: Blood group; sepsis; preterms
MeSH Terms: conditions — Premature Birth; Sepsis | interventions — Diagnosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- A blood group: prematurity with sepsis
  Interventions: Diagnostic Test: Diagnosis
- O blood group: prematurity with sepsis
  Interventions: Diagnostic Test: Diagnosis
- B blood group: prematurity with sepsis
  Interventions: Diagnostic Test: Diagnosis
- AB blood group: prematurity with sepsis
  Interventions: Diagnostic Test: Diagnosis

INTERVENTIONS:
Diagnostic Test: Diagnosis — biochemistry

SUMMARY:
To investigate whether there is a relationship between sepsis and blood groups in preterm infants.This retrospective cohort study included preterm neonates born at <32 weeks of gestation with a birth weight <1500 g. Neonates were grouped by blood type (O, A, B, AB) and sepsis were compared among these groups.

DETAILED DESCRIPTION:
This retrospective study was conducted on data collected between 1 January 2011 and 31 August 2018 in the neonatal intensive care unit (NICU) of the Health Sciences University Zekai Tahir Burak Women's Health Education and Research Hospital.

Neonates born at GA <32 weeks with birth weight (BW) <1500 g were included in the study.

Data pertaining to the neonates were recorded from medical records for each patient, and their ABO blood type was recorded.

The neonates were grouped by blood type (O, A, B, AB) and also separated into non-O (A, B, AB) and O groups and non-A (O, B, AB) and A groups for comparison of early and late onset sepsis.

ELIGIBILITY:
Inclusion Criteria:

* Preterm neonates born at <32 weeks of gestation with a birth weight <1500 g.

Exclusion Criteria:

* Neonates born with severe congenital defects, birth weight ≥1500 g and gestational age ≥32 weeks were excluded.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Neonates born at gestational age <32 weeks with birth weight <1500
Sampling Method: Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2018-12-15 (Estimated); Primary Completion 2019-02-01 (Estimated); Study Completion 2019-10-31 (Estimated)

PRIMARY OUTCOMES:
Association Between Different Blood Groups and Sepsis in Preterm Infants | Through study completion, an average of 3 month
  The neonates were grouped by blood type (O, A, B, AB) and also separated into non-O (A, B, AB) and O groups and non-A (O, B, AB) and A groups for comparison of demographic characteristics, clinical features, and sepsis.

CONTACTS AND LOCATIONS:
Overall Officials: ufuk cakir, Principal Investigator — Zekai Tahir Burak Women's Health Research and Education Hospital
Locations (1):
- Zekai Tahir Burak Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No